CLINICAL TRIAL: NCT06537167
Title: The Antihypertensive Effects of Transcutaneous Electrical Acupoint Stimulation in Patients With High-normal Blood Pressure and Grade 1 Hypertension
Brief Title: Transcutaneous Electrical Acupoint Stimulation on Blood Pressure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Institute of Hypertension (Other); Shanghai Jiao Tong University School of Biomedical engineering (Unknown)
Responsible Party: Principal Investigator, Ji-Guang Wang, Professor of the Shanghai Institute of Hypertension and the Department of Hypertension, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TEAS-BP
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: At the time of enrollment, each participant will be assigned a unique identification number (e.g., 001). The coded information will be stored in a secure database accessible only to designated members of the research team. A random number table will be generated using SPSS software, and participants will be allocated to either the "stimulation" experimental group or the "sham stimulation" control group according to the generated random numbers. Randomization information will be strictly confidential, ensuring that participants, outcome assessors, and statistical analysts are all blinded to the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "Stimulation" Experimental Group (Experimental)
  Interventions: Device: Transcutaneous electrical acupoint stimulation
- "Sham Stimulation" Control Group (Sham Comparator)
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Transcutaneous electrical acupoint stimulation — Participants will receive proper transcutaneous electrical acupoint stimulation treatment for three consecutive days. Each day, the selected five target acupoints (Renying, Quchi, Taichong, Zusanli, and Hegu) will be stimulated in rotation. Each acupoint will be stimulated once a day for 10 minutes, with a 2-minute interval between each acupoint, totaling 60 minutes. Throughout the trial, the stimulation parameters for each participant will remain constant, and the treatment will begin between 8:00 and 10:00 AM each day.
  Arms: "Stimulation" Experimental Group
Device: Sham stimulation — Participants will receive sham stimulation treatment, where the left-side skin near the selected five target acupoints (avoiding other functional acupoints) will be stimulated in rotation. The stimulation time and method will be the same as in the experimental group. Throughout the trial, the stimulation parameters for each participant will remain constant, and the treatment will begin between 8:00 and 10:00 AM each day.
  Arms: "Sham Stimulation" Control Group

SUMMARY:
This study will be conducted in patients with high-normal blood pressure and grade 1 hypertension and will be divided into two phases.

In Phase One, a small group of patients will undergo transcutaneous electrical acupoint stimulation treatment for three consecutive days. Blood pressure changes will be observed before and after each stimulation session, as well as 1 hour, 3 hours, and 5 hours after stimulation, during the night of the treatment day, and the next morning.

Phase Two will be a single-center, single-blind, parallel randomized controlled trial. After screening, patients will be randomly assigned to either the "stimulation" experimental group or the "sham stimulation" control group. For three consecutive days, both groups will receive their respective interventions at the same time each day, and their blood pressure changes will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Office systolic blood pressure between 130-150 mmHg and/or diastolic blood pressure between 80-95 mmHg
* Age between 18 and 75 years
* Not currently receiving antihypertensive medication or having discontinued antihypertensive medication for more than two weeks
* Able to undergo and complete the transcutaneous electrical acupoint stimulation treatment
* Agree to participate and sign the informed consent form

Exclusion Criteria:

* Pregnant or breastfeeding women
* Severe heart conditions, including coronary heart disease, myocardial infarction, arrhythmia, heart failure, or having an implanted cardiac pacemaker
* Skin conditions, including eczema, allergic dermatitis, or seborrheic dermatitis
* Neuromuscular diseases, mental disorders, epilepsy, or cognitive impairment
* Lower limb deep vein thrombosis or thrombophlebitis
* Wounds, surgical scars, or malignant tumors at the stimulation areas
* Inability to tolerate the transcutaneous electrical acupoint stimulation treatment or allergic to electrical stimulation
* Currently participating in other clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in office systolic blood pressure between the third day after TEAS treatment and the baseline (before the start of treatment on the first day) | At the third day after TEAS treatment and the baseline (before the start of treatment on the first day)

SECONDARY OUTCOMES:
Changes in office systolic blood pressure at other time points before and after treatment | At all other time points (excluding the third day after treatment) and the baseline (before the start of treatment on the first day)
Changes in office diastolic blood pressure at various time points before and after treatment | At each time point before and after treatment and the baseline (before the start of treatment on the first day).
Changes in ambulatory blood pressure before and after treatment | At the third day after the end of treatment and the baseline (before the start of treatment on the first day)
Changes in Hamilton Scale scores before and after treatment | At the third day after the end of treatment and the baseline (before the start of treatment on the first day)

IPD SHARING:
Plan to Share IPD: No